CLINICAL TRIAL: NCT02355275
Title: Thera-Band® Based Home Exercise Program for Low Back Pain Secondary Prevention
Brief Title: Thera-Band® HEP for LBP Secondary Prevention
Acronym: TBKT_HEP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: large non-response rate
Sponsor: Sport and Spine Rehab Clinical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SSR05
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Results first posted 2016-02-09 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-01

CONDITIONS: Low Back Pain
Keywords: Home Exercise; Resistance Exercise
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Home Exercise Program (Experimental)
  Interventions: Procedure: Home Exercise Program

INTERVENTIONS:
Procedure: Home Exercise Program — All patients will be provided with a Thera-Band® Loop and Band and handout describing home exercises to be performed 3 times a week for 4 weeks.

SUMMARY:
The purpose of this study is to determine the effectiveness of a Thera-Band based home exercise program (HEP) on LBP and disability 4 weeks post treatment discharge.

DETAILED DESCRIPTION:
The effectiveness of interventions for the treatment of acute and chronic LBP has been extensively studied, but study of the strategies for preventing the progression of acute LBP episodes into chronic back pain is still lacking. Therefore, determining the most effective secondary prevention strategy for the prevention of recurrences of LBP is essential for the reduction of long term disability. The purpose of this study is to determine the effectiveness of a Thera-Band based home exercise program (HEP) on LBP and disability 4 weeks post treatment discharge. A convenience sample of 22 new patients, 18-65 years of age, with current, chronic LBP will be recruited for this study at the discharge visit from care. Exclusionary criteria will include, current pregnancy and the presence of any red flags such as tumor or cancer, vertebral fracture, or infection. Upon agreeing to the study, patients will sign an informed consent, complete a demographics questionnaire, and complete specific outcome measure assessments. The outcome measures will include Numeric Pain Rating Scale (NPRS) and Oswestry Disability Index (ODI). Additionally, subjects will be asked to complete a secondary prevention program questionnaire. Following the initial paperwork, all patients will be provided with a Thera-Band® Loop and Band and handout describing the HEP to be performed 3 times a week for 4 weeks. At the conclusion of 4 weeks, a follow-up phone call or email, based on patient preference, will be conducted. The follow-up will include pain, disability, compliance, satisfaction of program of the home program.

ELIGIBILITY:
Inclusion Criteria:

* current, chronic low back pain
* discharging from care

Exclusion Criteria:

* current pregnancy
* presence of any red flags such as tumor or cancer, vertebral fracture, or infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sport & Spine Rehab, Rockville, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Home Exercise Program
Started | 22
Completed | 14
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Home Exercise Program
Number analyzed (Participants) | 22
Age, Continuous [Mean (Full Range); unit: years] | 41.5 [24 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Oswestry Disability Index
Description: Patient disability was measured using the Oswestry Disability Index (OSW), a self-report outcome measure. For each section the total possible score is 5: if the first statement is marked the section score = 0; if the last statement is marked, it = 5. The score is calculated by totaling the values marked, divided by 50 x 100. The greater the score the greater the disability. For example, 0% to 20% would be minimal disability and 81%-100% would be bed-bound. This outcome measure was reported at baseline (T1) and 4 weeks later (T2).
Time Frame: 4 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Home Exercise Program
Number analyzed (Participants) | 22
units on a scale
  OSW T1 | 18.75 [2 to 34]
  OSW T2 | 14.71 [4 to 42]

2. Secondary Outcome: Numeric Pain Rating Scale
Description: The Numeric Pain Rating Scale (NPRS) is a self-report scale measuring pain. It is measured from 0 to 10, 0 being pain free and 10 being the worse imaginable pain. This was measured at baseline (T1) and 4 weeks (T2)
Time Frame: 4 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Home Exercise Program
Number analyzed (Participants) | 22
units on a scale
  Pain T1 | 2.7 [0 to 7]
  Pain T2 | 2.3 [1 to 7]

ADVERSE EVENTS:
Arm/Group | Home Exercise Program
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No